CLINICAL TRIAL: NCT00027040
Title: HIV-Associated Cognitive Impairment and Oxidative Stress: An In Vivo Proton Magnetic Resonance Spectroscopy Study of Cerebral Injury
Brief Title: A Study of Decreased Mental Function Associated With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5114s; AACTG A5114s; ACTG A5114s
Record Dates: First submitted 2001-11-16; First posted 2001-11-19 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2012-10

CONDITIONS: Cognitive Disorders; HIV Infections
Keywords: AIDS Dementia Complex; Selegiline; Oxidative Stress; Cognition; Neuroprotective Agents; Brain Injuries; Magnetic Resonance Spectroscopy; Protons
MeSH Terms: conditions — Cognitive Dysfunction; HIV Infections; AIDS Dementia Complex; Brain Injuries | interventions — Selegiline

INTERVENTIONS:
Drug: Selegiline hydrochloride

SUMMARY:
The purpose of this study is to compare pictures of the brain of HIV-infected people with memory problems before and after treatment with selegiline. Selegiline is the study drug received through A5090.

HIV patients generally develop memory problems late in the disease. This will be examined using noninvasive proton magnetic resonance spectroscopy (1H-MRS). The effect of the drug selegiline on memory problems also will be examined.

DETAILED DESCRIPTION:
HIV-associated cognitive impairment generally develops during the later stages of the disease. This study proposes to non-invasively examine the pattern and extent of cerebral injury associated with HIV infection and its response to selegiline by using 1H-MRS. The following hypotheses will be tested: selegiline, a compound with antioxidant and anti-apoptotic properties, will reverse the metabolic abnormalities measured by 1H-MRS, and these changes will parallel the degree of improvement in cognitive and functional performance.

This is a substudy of ACTG A5090. The pattern and extent of cerebral injury associated with HIV infection and its response to selegiline are examined using a 1H-MRS. 1H-MRS evaluations are performed at screening and Week 24 (or at the time of premature discontinuation) of Step 1 of A5090. The screening MRS exams may only be performed once all A5090 screening evaluations (including the lumbar puncture) have been completed and it has been determined that the patient is eligible for A5090 study entry.

The screening MRS must be performed prior to A5090 study drug administration. The Week-24 MRS must be performed while the patient is still on blinded study drug.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are enrolled in ACTG protocol A5090.
* Meet the inclusion/exclusion criteria set forth for the Step 1 phase of AACTG protocol A5090.

Exclusion Criteria

Patients will not be eligible for this study if they have:

* Claustrophobia (unless sedation with lorazepam or zolpidem allows for safe performance of the MRS).
* Metallic implants/medical devices (e.g., skull implants or cardiac devices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Schifitto, Study Chair; Bradford Navia, Study Chair
Locations (12):
- United States (12):
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of California, San Diego, San Diego, California
  - Stanford University, Stanford, California
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hosp, Providence, Rhode Island
  - Stanley Street Treatment and Resource, Providence, Rhode Island
  - The Miriam Hosp, Providence, Rhode Island
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Result] Schifitto G, Yiannoutsos CT, Ernst T, Navia BA, Nath A, Sacktor N, Anderson C, Marra CM, Clifford DB; ACTG 5114 Team. Selegiline and oxidative stress in HIV-associated cognitive impairment. Neurology. 2009 Dec 8;73(23):1975-81. doi: 10.1212/WNL.0b013e3181c51a48. Epub 2009 Nov 4. PMID 19890073